CLINICAL TRIAL: NCT04916847
Title: Comparative Analysis of Anti-SARS-CoV-2 (Severe Acute Respiratory Syndrome) Humoral and Memory T Cell Responses in Children With Various Degrees of Immunosuppression: a Case-control Study
Brief Title: Comparative Analysis of Anti-COVID-19 (Severe Acute Respiratory Syndrome) Humoral and Memory T Cell Responses in Children With Various Degrees of Immunosuppression:
Acronym: PEDIMMCO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APH210217
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Immune Response
Keywords: children; SARS-CoV-2; Immunosuppression
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- children with controlled HIV: Children over 0 days and under 16 years old, with controlled HIV
  Interventions: Other: blood collection
- children with hematologic Malignancy treated by conventional chemotherapy: Children over 0 days and under 16 years old, with Hematologic Malignancy treated by conventional chemotherapy
  Interventions: Other: blood collection
- Children with inflammatory bowel disease treated by anti-TNF at least 6 weeks: Children over 0 days and under 16 years old, with inflammatory bowel disease treated by anti-TNF
  Interventions: Other: blood collection
- Children with idiopathic juvenile arthritis: Children over 0 days and under 16 years old, with idiopathic juvenile arthritis treated by methotrexate:
  Interventions: Other: blood collection
- Children treated by renal transplantation: Children over 0 days and under 16 years old, treated by renal transplantation from more than 3 months:
  Interventions: Other: blood collection
- Children attending consultation: Children over 0 days and under 16 years old, without immunodepression or chronic inflammation attending consultation for :
  * preoperative assessment
  * -congenital abnormalities of the kidney and urinary tract:
  * Nephropathies without renal impairment (eDFG > 45mL/min/1.73m2)
  * Non-inflammatory intestinal (polyposis, Chronic intestinal pseudo-obstruction, short bowel syndrome) or pancreatic (hereditary pancreatitis) pathologies This group of children will be a control group (age matched healthy children, non-immunosuppressed).
  Interventions: Other: blood collection

INTERVENTIONS:
Other: blood collection — Depending on the weight of the child, between 5ml and 15ml of blood will be collected during a blood test necessary for the conventional care of the patient. A second blood sample will be taken one year later. The volume of blood taken does not exceed the volume allowed by the guideline "Ethical considerations for clinical trials of medicinal products conducted in the paediatric population".
  We will analyse:
  1. Specific antibody responses (IgM, IgG, and immunoglobulin A (IgA) anti SARS-Cov-2) by quantitative chemiluminescence analysis.
  2. Protective neutralizing capacity of these antibodies (neutralizing antibodies against SARS-cOV-2) by neutralization test.
  3. SARS-Cov-2 specific memory T cell responses by multiparametric flow cytometry in order to characterize their maturation, differentiation, senescence, activation, secretion of interleukin (cytokines 2) , IFN-g, TNF) or Interferon-gamma (IFN-g) ELISPOT assay.

SUMMARY:
Adaptive immune responses are essential for clearing viral infections and retention of virus specific memory populations is required for long-term immunity. However, there is still uncertainty about whether adaptive immune responses to SARS-CoV-2 are protective. Such knowledge is of immediate relevance, as it will provide insights into immunity of SARS-CoV-2 infection and thus help define future immunization strategies. Because of the importance of asymptomatic cases in children, a specific study is needed in this population in order to determine their individual and collective protective capacity. This is even truer for immune compromised children that likely have severe forms of the disease with active and prolonged viral replication in whom it is therefore essential to determine the extent of sero conversion but also the quality and duration of the memory responses.

For this purpose, we plan to analyze the anti-SARS-CoV-2 humoral and memory T cell responses, in different groups of immuno-compromized children (i.e with different levels/type of immunosuppression; HIV, renal or stem cell transplantation, anti-TNF or methotrexate treatment) and healthy controls seen in 3 University Hospitals, in order to determine the proportion of children with SARS-CoV-2 specific humoral responses, their protective capacity, the magnitude and the quality of the SARS-Cov-2 memory T cells but also their long term persistence at 1 year.

DETAILED DESCRIPTION:
Adaptive immune responses are essential for clearing viral infections and retention of virus specific memory populations is required for long-term immunity. However, there is still uncertainty about whether adaptive immune responses to SARS-CoV-2 are protective. Such knowledge is of immediate relevance, as it will provide insights into immunity of SARS-CoV-2 infection and thus help define future immunization strategies. Because of the importance of asymptomatic cases in children, a specific study is needed in this population in order to determine their individual and collective protective capacity. This is even truer for immuno-compromised children that likely have severe forms of the disease with active and prolonged viral replication in whom it is therefore essential to determine the extent of seroconversion but also the quality and duration of the memory responses.

For this purpose, we plan to analyze the anti-SARS-CoV-2 humoral and memory T cell responses, in different groups of immuno-compromized children (i.e with different levels/type of immunosuppression; HIV, renal or stem cell transplantation, anti-TNF or methotrexate treatment) and healthy controls seen in 3 University Hospitals, in order to determine the proportion of children with SARS-CoV-2 specific humoral responses, their protective capacity, the magnitude and the quality of the SARS-Cov-2 memory T cells but also their long term persistence at 1 year.

In this study, we will evaluate the proportion of children who developed anti-SARS-CoV-2 humoral and cellular memory immune responses and the protective capacity of these responses in different groups of immune-compromised children.

As explained above, clinical significance of SARS-CoV-2 varies among different immune-compromised populations, in relation to the individual degree and type of immunosuppression. It is therefore necessary to obtain data on post infection protective immunity in different groups of immunosuppressed children. The intervention added for this study, blood samples will be taken. The blood sample will consist of two to three (depending on weight) additional tubes (heparin-lithium, dry) between 5 ml and 15 ml each taken during a blood test necessary for the patient's standard care. A second blood sample will be taken one year later for those with a positive response to SARS-CoV-2 and for vaccinated children. The volume of blood taken does not exceed the volume allowed by the guideline "Ethical considerations for clinical trials of drugs in the pediatric population".

ELIGIBILITY:
Inclusion Criteria:

* Children over 0 days and under 16 years of age seen in consultation for the follow-up of their pathology or immunosuppressive treatment (see above, Groups of patients).
* Several cases groups will be considered in this study, presented with immunocompromised state or immunosuppressive treatment (i. e. children with: HIV infection, Hematologic Malignancy treated by conventional chemotherapy, Hematologic pathology treated by allogenic stem cell transplantation, inflammatory bowel disease treated by anti-TNF, idiopathic juvenile arthritis treated by methotrexate, treated by renal transplantation; see above, paragraph groups of patients for details).

Children over 0 days and under 16 years of age considered as control will be non-immunosuppressed children without chronic inflammation, attending consultation for preoperative assessment or congenital abnormalities of the kidney and urinary tract, for Nephropathies without renal impairment (eDFG > 45mL/min/1.73m), for non-inflammatory intestinal (polyposis, Chronic intestinal pseudo-obstruction, short bowel syndrome) or pancreatic (hereditary pancreatitis) pathologies.For comparisons, healthy children will be age-matched with each case.

* Informed consent of the holder (s) of the exercise of parental authority
* Affiliation to a social security scheme

Exclusion Criteria:

* Children who have a signs of a current infection.
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* Children who received one or more doses of SARS-Cov-2 vaccine.

Ages: 1 Day to 15 Years | Sex: All
Age Groups: Child
Study Population: In this study, we will evaluate the proportion of children who developed anti-SARS-CoV-2 humoral and cellular memory immune responses and the protective capacity of these responses in different groups of immune-compromised children.
  As explained above, clinical significance of SARS-CoV-2 varies among different immune-compromised populations, in relation to the individual degree and type of immunosuppression. It is therefore necessary to obtain data on post infection protective immunity in different groups of immunosuppressed children.
  To these purpose, the study will benefit from a Network of Pediatric Physicians used to work or collaborating together, with experience of children's studies and strong adherence to the study.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Numbers of subjects with positive IgM | at baseline
  Numbers of subjects with positive IgM titer levels against SARS-Cov-2 (according to the manufacturer) at baseline.

SECONDARY OUTCOMES:
Numbers of subjects with positive IgG | at baseline and at 12 months
  Numbers of subjects with positive immunoglobulin G (IgG) SARS-Cov-2 (according to the manufacturer)
Numbers of subjects with positive titers | at baseline and at 12 months
  Number of subjects with positive titers
Percentage of SARS-CoV-2 memory T | at baseline ans at 12 months
  Percentage and counts of SARS-CoV-2 memory T cells in lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Carcelain Guislaine, PhD, Study Chair — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France